CLINICAL TRIAL: NCT00129064
Title: Improving the Outpatient Referral Process With Electronic Communications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Commonwealth Fund (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2004-P-000710; 20010373
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Communication; Interprofessional Relations
Keywords: Referrals; Quality of care; Ambulatory care; Electronic medical record; Referral communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Electronic referral system

SUMMARY:
An electronic referral application will be developed and integrated into the existing outpatient information system. The primary goal of this software is to improve the quality and coordination of patient care by increasing physician-to-physician communication. The investigators anticipate that improved communications will also enhance physician and patient satisfaction and provide cost savings. These outcomes will be formally evaluated following implementation of the application.

DETAILED DESCRIPTION:
A trial will be performed to test and quantify the benefits of electronic referrals. Primary care physicians (PCPs) from 2 community-based clinics will be recruited for enrollment. The control group will initiate referrals using the pre-existing paper forms; physician-to-physician communication can occur by e-mail, phone, or mail at the discretion of the referring physician as is currently the standard. Physicians randomized to the intervention arm will be asked to use the electronic application for every referral during the study period. For 6 months, every new referral initiated within the study groups will be assessed for the completeness of patient information and timing of feedback to the referring physician via physician surveys. In addition, a subgroup of patients in the control and intervention arms will be surveyed to assess the impact of the intervention on patient satisfaction with the referral process.

ELIGIBILITY:
Inclusion Criteria:

* Any referral initiated by a PCP at the study sites for a patient to go to a specialist for the first time

Exclusion Criteria:

* Referrals for repeat specialist visits or referrals not initiated by a PCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-11; Study Completion 2007-03

PRIMARY OUTCOMES:
Percentage of referral requests with complete information
Percentage of referrals with timely information exchanged

SECONDARY OUTCOMES:
Physician satisfaction
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Tejal K Gandhi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's, Boston, Massachusetts, United States